CLINICAL TRIAL: NCT01872533
Title: Effect of 10-day Overnight Hypoxia Treatment on Whole Body Insulin Sensitivity (SLEEP HIGH Study)
Acronym: SLEEP HIGH
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Eric Ravussin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PBRC 11009
Record Dates: First submitted 2013-06-03; First posted 2013-06-07 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Insulin Resistance
Keywords: obesity; hypoxia; insulin sensitivity; altitude
MeSH Terms: conditions — Insulin Resistance; Obesity; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypoxia Exposure (Experimental): There was only one study arm: All participants slept in moderate hypoxia (see description below).
  Interventions: Other: Hypoxia Exposure

INTERVENTIONS:
Other: Hypoxia Exposure — Participants spent 10 consecutive nights (approximately 100 hours of exposure) in a hypoxic tent at ~ 15% O2 (ca. 2400 m elevation).

SUMMARY:
The purpose of this study is to look at how a reduction in oxygen levels (hypoxia) influences insulin sensitivity and carbohydrate metabolism. It is expected that 10 nights of exposure to moderate hypoxia (~ 15% O2, similar to conditions at an altitude of ~7500 feet) will improve glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-45 years
* Male
* Obese category (BMI > 30 kg/m2)
* Healthy as assessed by a self-reported health questionnaire
* Non-smokers
* Weight stable over the past 3 months (<2kg fluctuation)

Exclusion Criteria:

* Female
* Diabetes
* Sleep apnea
* Hypertension
* History of altitude sickness
* Individuals taking any chronic medications
* Individuals taking any stimulants
* Individuals taking beta-blockers
* Individuals with chronic alcohol consumption (>3 drinks per day) or drug abuse.
* Individuals unable to abstain from caffeinated beverage or alcohol the days of study testing
* Individuals with history disease or history of stroke

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in Insulin sensitivity | Change from baseline to 10 nights of hypoxia exposure
  Glucose disposal and oxidation were measured using a two-step hyperinsulinemic euglycemic clamp and indirect calorimetry.

SECONDARY OUTCOMES:
Change in oxygen tension in adipose tissue | Before and after 10 nights of hypoxia exposure
  pO2 levels were measured in adipose tissue both under hypoxia and normal oxygen conditions (normoxia) via a dual temperature-oxygen tension probe.
Glucose uptake in myotubes | Before 10 nights of hypoxia exposure
  Glucose uptake assays were performed in the presence or absence of hypoxia on myotubes harvested from muscle biopsies.
Change in gene and protein expression | Before and after 10 nights of hypoxia exposure
  Gene and protein expression of some hypoxia-responsive and insulin-signaling markers were measured in biopsied muscle and adipose tissue via RT-PCR and Western blotting, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Lecoultre V, Peterson CM, Covington JD, Ebenezer PJ, Frost EA, Schwarz JM, Ravussin E. Ten nights of moderate hypoxia improves insulin sensitivity in obese humans. Diabetes Care. 2013 Dec;36(12):e197-8. doi: 10.2337/dc13-1350. No abstract available. PMID 24265370